CLINICAL TRIAL: NCT03719365
Title: Driving Pressure Variation During Proportional Assisted Ventilation: Comparison Between NAVA and PSV
Brief Title: Driving Pressure Variation: NAVA vs PSV
Acronym: DPNAVA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Gianmaria Cammarota, Principal investigator, Azienda Ospedaliero Universitaria Maggiore della Carita
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CE 110/18
Record Dates: First submitted 2018-10-19; First posted 2018-10-25 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Mechanical Ventilation Complication; Ventilator-Induced Lung Injury
Keywords: PSV; NAVA; Driving Pressure; Mechanical Assisted Ventilation
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Intervention Model Description: Randomized, interventional, prospective study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NAVAPSV (Experimental): Each patient enrolled in the study will be submitted to 3 ventilation trials during PSV and NAVA ventilation modes, assigned in a randomized order.
  Interventions: Device: NAVAPSV

INTERVENTIONS:
Device: NAVAPSV — During the first trial, PSV will be set in order to obtain a Vt between 6 and 8 ml/kg; this support level will be defined as PSV100. Subsequently, the corresponding NAVA level (NAVA 100) will be determined using a dedicated ventilator function (NAVA Preview) which is able to estimate NAVA level in order to deliver an equivalent inspiratory peak pressure (Paw peak) compared to that obtained during PSV mode. Afterwards, PSV100 and NAVA100 will be first increased (PSV150 and NAVA150) during the second trial and then decreased during the third trial (PSV50 and NAVA150) by 50% from basal value. During the study period, PEEP and FiO2 will be kept equal to the values in use before patient enrollment.

SUMMARY:
Assisted ventilation represents, nowadays, the preferred ventilation mode in clinical practice.It has been shown that assisted ventilation modes improve ventilation/perfusion matching, descrease risk of Ventilator induced lung injury and muscle atrophy and have less influence on haemodynamic function.

However, PSV (Pressure Support Ventilation) is not free from complications: it may worsen or cause lung injuries by increasing alveolar and intrathoracic negative pressure and by loosing control on Tidal Volume (Vt). Indeed, it has been demonstrated that Vt is the main factor related to VILI.

It has been shown that lower Vt and higher PEEP can improve clinical outcome only if associated with a simultaneous reduction in Driving Pressure. Increase in Driving Pressure resulted strongly associated with negative outcomes, especially if higher than 15 cm H2O.

PSV is currently the most used assisted ventilation mode. NAVA (Neurally Adjusted Ventilatory Assist) is a ventilation mode in which the diaphragmatic electrical activity (EAdi) is used as a trigger to start a mechanical breath, applying positive pressure during patient's inspiration. Diaphragmatic electrical activity (EAdi) can be detected by a particular nasogastric tube (EAdi catheter). EAdi is the currently available signal closest to the neural breathing centers, which can estimate the patient's respiratory drive, if phrenic nerves are not damaged. It has been demonstrated that NAVA ventilation can reduce the incidence of patient-ventilator asynchronies, because the delivery of the support and the cycling between inspiration and expiration are completely controlled by the patient.

However, although PSV and NAVA have been widely compared in many investigations, up to now there are no studies about driving pressure variation during these two modalities of mechanical assisted ventilation. The aim of this study is to measure changes in driving pressure at different levels of ventilatory assistance in PSV and NAVA ventilation modes.

Secondary end points are respiratory mechanics indices and patient/ventilator related asynchrony evaluation and comparison.

DETAILED DESCRIPTION:
Any patient who is already on an assisted mode of ventilation and displays triggering efforts will be enrolled in the study and will be submitted to 3 ventilation trials, in PSV and NAVA ventilation modes; each trial will last 20 minutes. Every trial will be performed in a randomized order, based on random computer generated sequences.

During the first trial, PSV will be set in order to obtain a Vt between 6 and 8 ml/kg;this support level will be defined as PSV100. Subsequently, the corresponding NAVA level (NAVA 100) will be determined using a dedicated ventilator function (NAVA Preview) which is able to estimate NAVA level in order to deliver an equivalent inspiratory peak pressure (Paw peak) compared to that obtained during PSV mode. Afterwards, pressure support level of assistance of PSV100 and NAVA100 will be firstly increased (PSV150 and NAVA150) during the second trial and then decreased during the third trial (PSV50 and NAVA150) by 50% from basal value.

During the study period, PEEP and FiO2 will be kept equal to the values in use before patient enrollment. End-inspiration and end-expiration pauses will be performed at the end of each trial by pressing the dedicated button on the ventilator control panel. Airway pressure and flow will be recorded.

Patients, as usual, clinical practice, will be sedated at different levels and this could compromise their content of consciousness.

At the beginning of each trial, an endotracheal tube suction will be done. Last 5 minutes of each trial will be recorded and stored in a computer for subsequent statistical analysis. Respiratory mechanical indices (airway pressure, tidal volume, flow) and electric diaphragmatic activity will be recorded by a dedicated software called NAVA- tracker. At the end of each trial an arterial blood gas analysis (ABGs) will be performed to evaluate PaCO2, PH and blood oxygenation (PaO2). at the end of each trial, an ultrasound evaluation of diaphragm will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Every patients undergoing partial assisted mechanical ventilation

Exclusion Criteria:

* Gastro-esophageal surgery in the previous 12 months;
* Gastro-esophageal bleeding in the previous 30 days;
* Esophageal varices history;
* Maxillo-facial surgery or trauma;
* Haemodinamic instability despite adequate fluid infusion (i.e. need for continuous infusion epinephrine or vasopressin or dopamine at a dose greater than 5 mcg/kg/min to obtain systolic pressure > 90 mmHg);
* Body temperature > 38° C during the study screening;
* Coagulation disorders (INR > 1.5, aPTT > 44 sec);
* Vt < 8 ml/kg with minimum inspiratory effort of 8 cmH2O;
* Inclusion in other research protocols

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Driving pressure in PSV and NAVA | At the end of every 20 minutes lasting ventilation trial.
  Driving Pressure measurements in in PSV and NAVA (cmH2O)

SECONDARY OUTCOMES:
Respiratory mechanical indices variation | At the end of every 20 minutes lasting ventilation trial.
  electrical diaphragmatic activity (mcvolts)
Patient/ventilator interaction | At the end of every 20 minutes lasting ventilation trial.
  asynchrony index (normal value < 10%; pathological value > 10%)
Patient/ventilator interaction | At the end of every 20 minutes lasting ventilation trial.
  time of synchrony (msec)
diaphragm ultrasound | At the end of every 20 minutes lasting ventilation trial.
  evaluation of diaphragm performance at each trial

CONTACTS AND LOCATIONS:
Overall Officials: Gianmaria Cammarota, MD, PhD, Principal Investigator — AOU Maggiore della Carità
Locations (1):
- A.O.U Maggiore della Carità, Novara, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Putensen C, Zech S, Wrigge H, Zinserling J, Stuber F, Von Spiegel T, Mutz N. Long-term effects of spontaneous breathing during ventilatory support in patients with acute lung injury. Am J Respir Crit Care Med. 2001 Jul 1;164(1):43-9. doi: 10.1164/ajrccm.164.1.2001078. PMID 11435237
- [Background] Putensen C, Mutz NJ, Putensen-Himmer G, Zinserling J. Spontaneous breathing during ventilatory support improves ventilation-perfusion distributions in patients with acute respiratory distress syndrome. Am J Respir Crit Care Med. 1999 Apr;159(4 Pt 1):1241-8. doi: 10.1164/ajrccm.159.4.9806077. PMID 10194172
- [Background] Grasso F, Engelberts D, Helm E, Frndova H, Jarvis S, Talakoub O, McKerlie C, Babyn P, Post M, Kavanagh BP. Negative-pressure ventilation: better oxygenation and less lung injury. Am J Respir Crit Care Med. 2008 Feb 15;177(4):412-8. doi: 10.1164/rccm.200707-1004OC. Epub 2007 Dec 13. PMID 18079496
- [Background] Xia J, Zhang H, Sun B, Yang R, He H, Zhan Q. Spontaneous breathing with biphasic positive airway pressure attenuates lung injury in hydrochloric acid-induced acute respiratory distress syndrome. Anesthesiology. 2014 Jun;120(6):1441-9. doi: 10.1097/ALN.0000000000000259. PMID 24722174
- [Background] Futier E, Constantin JM, Combaret L, Mosoni L, Roszyk L, Sapin V, Attaix D, Jung B, Jaber S, Bazin JE. Pressure support ventilation attenuates ventilator-induced protein modifications in the diaphragm. Crit Care. 2008;12(5):R116. doi: 10.1186/cc7010. Epub 2008 Sep 11. PMID 18786263
- [Background] Yoshida T, Uchiyama A, Matsuura N, Mashimo T, Fujino Y. Spontaneous breathing during lung-protective ventilation in an experimental acute lung injury model: high transpulmonary pressure associated with strong spontaneous breathing effort may worsen lung injury. Crit Care Med. 2012 May;40(5):1578-85. doi: 10.1097/CCM.0b013e3182451c40. PMID 22430241
- [Background] Yoshida T, Torsani V, Gomes S, De Santis RR, Beraldo MA, Costa EL, Tucci MR, Zin WA, Kavanagh BP, Amato MB. Spontaneous effort causes occult pendelluft during mechanical ventilation. Am J Respir Crit Care Med. 2013 Dec 15;188(12):1420-7. doi: 10.1164/rccm.201303-0539OC. PMID 24199628
- [Background] Yoshida T, Uchiyama A, Matsuura N, Mashimo T, Fujino Y. The comparison of spontaneous breathing and muscle paralysis in two different severities of experimental lung injury. Crit Care Med. 2013 Feb;41(2):536-45. doi: 10.1097/CCM.0b013e3182711972. PMID 23263584
- [Background] Amato MB, Barbas CS, Medeiros DM, Magaldi RB, Schettino GP, Lorenzi-Filho G, Kairalla RA, Deheinzelin D, Munoz C, Oliveira R, Takagaki TY, Carvalho CR. Effect of a protective-ventilation strategy on mortality in the acute respiratory distress syndrome. N Engl J Med. 1998 Feb 5;338(6):347-54. doi: 10.1056/NEJM199802053380602. PMID 9449727
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Malhotra A. Low-tidal-volume ventilation in the acute respiratory distress syndrome. N Engl J Med. 2007 Sep 13;357(11):1113-20. doi: 10.1056/NEJMct074213. PMID 17855672
- [Background] Mascia L, Pasero D, Slutsky AS, Arguis MJ, Berardino M, Grasso S, Munari M, Boifava S, Cornara G, Della Corte F, Vivaldi N, Malacarne P, Del Gaudio P, Livigni S, Zavala E, Filippini C, Martin EL, Donadio PP, Mastromauro I, Ranieri VM. Effect of a lung protective strategy for organ donors on eligibility and availability of lungs for transplantation: a randomized controlled trial. JAMA. 2010 Dec 15;304(23):2620-7. doi: 10.1001/jama.2010.1796. PMID 21156950
- [Background] Serpa Neto A, Cardoso SO, Manetta JA, Pereira VG, Esposito DC, Pasqualucci Mde O, Damasceno MC, Schultz MJ. Association between use of lung-protective ventilation with lower tidal volumes and clinical outcomes among patients without acute respiratory distress syndrome: a meta-analysis. JAMA. 2012 Oct 24;308(16):1651-9. doi: 10.1001/jama.2012.13730. PMID 23093163
- [Background] Futier E, Constantin JM, Paugam-Burtz C, Pascal J, Eurin M, Neuschwander A, Marret E, Beaussier M, Gutton C, Lefrant JY, Allaouchiche B, Verzilli D, Leone M, De Jong A, Bazin JE, Pereira B, Jaber S; IMPROVE Study Group. A trial of intraoperative low-tidal-volume ventilation in abdominal surgery. N Engl J Med. 2013 Aug 1;369(5):428-37. doi: 10.1056/NEJMoa1301082. PMID 23902482
- [Background] Amato MB, Meade MO, Slutsky AS, Brochard L, Costa EL, Schoenfeld DA, Stewart TE, Briel M, Talmor D, Mercat A, Richard JC, Carvalho CR, Brower RG. Driving pressure and survival in the acute respiratory distress syndrome. N Engl J Med. 2015 Feb 19;372(8):747-55. doi: 10.1056/NEJMsa1410639. PMID 25693014
- [Background] MacIntyre NR. Respiratory function during pressure support ventilation. Chest. 1986 May;89(5):677-83. doi: 10.1378/chest.89.5.677. PMID 3698697
- [Background] Brochard L, Pluskwa F, Lemaire F. Improved efficacy of spontaneous breathing with inspiratory pressure support. Am Rev Respir Dis. 1987 Aug;136(2):411-5. doi: 10.1164/ajrccm/136.2.411. PMID 3619200
- [Background] Cereda M, Foti G, Marcora B, Gili M, Giacomini M, Sparacino ME, Pesenti A. Pressure support ventilation in patients with acute lung injury. Crit Care Med. 2000 May;28(5):1269-75. doi: 10.1097/00003246-200005000-00002. PMID 10834664
- [Background] Nava S, Bruschi C, Fracchia C, Braschi A, Rubini F. Patient-ventilator interaction and inspiratory effort during pressure support ventilation in patients with different pathologies. Eur Respir J. 1997 Jan;10(1):177-83. doi: 10.1183/09031936.97.10010177. PMID 9032512
- [Background] Esteban A, Anzueto A, Alia I, Gordo F, Apezteguia C, Palizas F, Cide D, Goldwaser R, Soto L, Bugedo G, Rodrigo C, Pimentel J, Raimondi G, Tobin MJ. How is mechanical ventilation employed in the intensive care unit? An international utilization review. Am J Respir Crit Care Med. 2000 May;161(5):1450-8. doi: 10.1164/ajrccm.161.5.9902018. PMID 10806138
- [Background] Spahija J, de Marchie M, Albert M, Bellemare P, Delisle S, Beck J, Sinderby C. Patient-ventilator interaction during pressure support ventilation and neurally adjusted ventilatory assist. Crit Care Med. 2010 Feb;38(2):518-26. doi: 10.1097/CCM.0b013e3181cb0d7b. PMID 20083921
- [Background] Ferreira JC, Diniz-Silva F, Moriya HT, Alencar AM, Amato MBP, Carvalho CRR. Neurally Adjusted Ventilatory Assist (NAVA) or Pressure Support Ventilation (PSV) during spontaneous breathing trials in critically ill patients: a crossover trial. BMC Pulm Med. 2017 Nov 7;17(1):139. doi: 10.1186/s12890-017-0484-5. PMID 29115949
- [Background] Sinderby C, Beck J, Spahija J, de Marchie M, Lacroix J, Navalesi P, Slutsky AS. Inspiratory muscle unloading by neurally adjusted ventilatory assist during maximal inspiratory efforts in healthy subjects. Chest. 2007 Mar;131(3):711-717. doi: 10.1378/chest.06-1909. PMID 17356084
- [Derived] Cammarota G, Verdina F, De Vita N, Boniolo E, Tarquini R, Messina A, Zanoni M, Navalesi P, Vetrugno L, Bignami E, Corte FD, De Robertis E, Santangelo E, Vaschetto R. Effects of Varying Levels of Inspiratory Assistance with Pressure Support Ventilation and Neurally Adjusted Ventilatory Assist on Driving Pressure in Patients Recovering from Hypoxemic Respiratory Failure. J Clin Monit Comput. 2022 Apr;36(2):419-427. doi: 10.1007/s10877-021-00668-2. Epub 2021 Feb 9. PMID 33559864